CLINICAL TRIAL: NCT01357109
Title: Effect of Bosentan on Macro- and Microvascular Function in Patients With Type 2 Diabetes
Brief Title: Effect of Bosentan on Endothelial Function in Patients With Type 2 Diabetes
Acronym: BANDY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Swedish Heart Lung Foundation (Other); The Swedish Research Council (Other Government); Actelion (Industry)
Responsible Party: John Pernow, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BANDY 070112; 2007-000221-22 (EudraCT Number)
Record Dates: First submitted 2011-05-18; First posted 2011-05-20 (Estimated); Last update posted 2011-05-20 (Estimated); Status verified 2007-10

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Bosentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bosentan (Experimental)
  Interventions: Drug: Bosentan
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bosentan — 62.5 mg bid for two weeks and 125 mg bid for two weeks
  Arms: Bosentan
Drug: Placebo — Matched placebo bid
  Arms: Placebo

SUMMARY:
The purpose of the study is to investigate if oral treatment with bosentan improves endothelium-dependent vasodilatation in patients with type 2 diabetes and microangiopathy.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetes mellitus type 2 of >2 years duration
2. Albuminuria

Exclusion Criteria:

1. Age >80 years
2. Myocardial infarction/unstable angina within three months prior to randomisation
3. Decompensated congestive heart failure or functional class 3 and 4.
4. Changes in dosage of any vasodilator drugs during the preceding six weeks
5. Women of fertile age.
6. Impaired hepatic function (2 times upper normal limit of aminotransferases ASAT and ALAT)
7. Ongoing treatment with glibenclamide, cyclosporin or warfarin
8. Any concomitant disease or condition that may interfere with the possibility for the patient to comply with or complete the study protocol
9. Participant in an ongoing study
10. Unwillingness to participate following oral and written information

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-11; Primary Completion 2010-04 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Peripheral endothelial function | 4 weeks

SECONDARY OUTCOMES:
Inflammatory markers | 4 weeks
Renal protein excretion | 4 weeks
Myocardial perfusion | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John Pernow, Dr, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Rafnsson A, Bohm F, Settergren M, Gonon A, Brismar K, Pernow J. The endothelin receptor antagonist bosentan improves peripheral endothelial function in patients with type 2 diabetes mellitus and microalbuminuria: a randomised trial. Diabetologia. 2012 Mar;55(3):600-7. doi: 10.1007/s00125-011-2415-y. Epub 2011 Dec 27. PMID 22200728